CLINICAL TRIAL: NCT02296892
Title: A Phase III Study Evaluating the Efficacy and Safety of Remimazolam (CNS 7056) Compared to Placebo and Midazolam in Patients Undergoing Bronchoscopy
Brief Title: A Phase III Study of Remimazolam in Patients Undergoing Bronchoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Paion UK Ltd. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNS7056-008
Record Dates: First submitted 2014-11-11; First posted 2014-11-21 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Bronchoscopy
Keywords: Remimazolam, midazolam, bronchoscopy, procedural sedation
MeSH Terms: interventions — remimazolam; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Remimazolam (Experimental): Double-blind Remimazolam arm: 5 mg iv for sedation induction, and 2.5 mg iv top-ups for sedation maintenance.
  Fentanyl pre-treatment: 25-50 μg (or less for elderly/disabled subjects), and 25 μg top-up doses
  Interventions: Drug: Remimazolam
- Placebo (Placebo Comparator): Double-blind placebo arm as inactive control
  Fentanyl pre-treatment: 25-50 μg (or less for elderly/disabled subjects), and 25 μg top-up doses
  Interventions: Drug: Placebo
- Midazolam (Active Comparator): Open-label Midazolam arm: 1.75 mg* iv for sedation induction and 1.0 mg* iv for sedation maintenance. *1.0 mg for induction and 0.5 mg for maintenance in adults over 60, debilitated or chronically ill.
  Fentanyl pre-treatment: 25-50 μg (or less for elderly/disabled subjects), and 25 μg top-up doses
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Remimazolam — For induction and maintenance of sedation
  Other Names: CNS7056
  Arms: Remimazolam
Drug: Placebo — Inactive control arm
  Arms: Placebo
Drug: Midazolam — For induction and maintenance of sedation
  Other Names: Versed
  Arms: Midazolam

SUMMARY:
A prospective, double-blind, randomized, placebo and active controlled, multi-center, parallel group study comparing remimazolam to placebo, with an additional open label arm for midazolam, in patients undergoing a bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, aged ≥18 years, scheduled to undergo a diagnostic or therapeutic flexible bronchoscopy in the bronchoscopy suite (therapeutic bronchoscopies could include eg, lavage, biopsies, brushings, and foreign body extraction).
2. American Society of Anesthesiologists Physical Status Score (ASA PS) 1 through 3.
3. Body mass index (BMI) ≤ 45.
4. Peripheral blood oxygen saturation (measured by pulse oximetry: SpO2) ≥ 90% in ambient air or with no more than 2 L/min of oxygen support.
5. For all female patients, negative result of urine pregnancy test. Additionally, for women of child bearing potential only, use of birth control during the study period (from the time of consent until all specified observations were completed).
6. Patients voluntarily signed and dated an informed consent form that was approved by an IRB prior to the conduct of any study procedure, including screening procedures.
7. Patient was willing and able to comply with study requirements and available for a follow up phone call on Day Day 4 (+3/ 1 days) after the bronchoscopy.

Exclusion Criteria:

1. Patients with a known sensitivity to benzodiazepines, flumazenil, opioids, naloxone, or a medical condition such that these agents were contraindicated.
2. Bronchoscopy outside the bronchoscopy unit (eg, intensive care unit).
3. Patients on mechanical ventilation.
4. Tracheal stenosis.
5. Planned laser bronchoscopy, rigid scope bronchoscopy.
6. Use of unstable doses of benzodiazepines and opioids for any indication, eg, insomnia, anxiety, or spasticity. An unstable dose means dose changes of more than 50% of the previous dose within 30 days prior to Day of procedure.
7. Female patients with a positive pregnancy test at Screening or Baseline and lactating female patients.
8. Patients with positive drugs of abuse screen (unless explained by concomitant medication) or a positive ethanol test at baseline.
9. Patient with a history of drug or ethanol abuse within the past two years.
10. Patients in receipt of any investigational drug or use of investigational device within 30 days or less than 7 t½ (whichever was longer) before the start of the study or scheduled to receive one during the study period.
11. Participation in any previous clinical study with remimazolam.
12. Patients with an inability to communicate well in English with the investigator or deemed unsuitable according to the investigator (in each case providing a reason).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Silvestri, MD, Principal Investigator — Medical University of South Carolina, US
Locations (14):
- United States (14):
  - Pab Clinical Research, Brandon, Florida
  - Sun City Office, Sun City Center, Florida
  - Laporte County Institute For Clinical Research, Michigan City, Indiana
  - The Johns Hopkins Center for Interventional and Pulmonary Care, Baltimore, Maryland
  - Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri
  - Unc Division of Pulmonary and Critical Care, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - S. Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - Pulmonary Associates of Richmond, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Multicare Institute For Research & Innovation, Tacoma, Washington

REFERENCES:
- [Result] Pastis NJ, Yarmus LB, Schippers F, Ostroff R, Chen A, Akulian J, Wahidi M, Shojaee S, Tanner NT, Callahan SP, Feldman G, Lorch DG Jr, Ndukwu I, Pritchett MA, Silvestri GA; PAION Investigators. Safety and Efficacy of Remimazolam Compared With Placebo and Midazolam for Moderate Sedation During Bronchoscopy. Chest. 2019 Jan;155(1):137-146. doi: 10.1016/j.chest.2018.09.015. Epub 2018 Oct 4. PMID 30292760

RESULTS

PARTICIPANT FLOW:
Groups:
- Remimazolam: Remimazolam iv 5 mg for sedation induction, and 2.5 mg top-ups for sedation maintenance.
- Placebo: Placebo iv as inactive control arm
- Midazolam: Midazolam iv 1.75 mg* for sedation induction and 1.0 mg* for sedation maintenance. *1.0 mg for induction and 0.5 mg for maintenance in adults over 60, debilitated or chronically ill.
Period: Overall Study
Arm/Group | Remimazolam | Placebo | Midazolam
Started | 310 | 63 | 73
Safety Population (All randomized patients who received any amount of the trial drug and were analyzed as treated) | 303 | 59 | 69
Complete Trial Treatment Period | 303 | 59 | 69
Completed | 298 | 59 | 68
Not Completed | 12 | 4 | 5
Not completed — Exclusion Criteria at Day of Procedure | 7 | 4 | 4
Not completed — Lost to Follow-up | 5 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population is the Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Remimazolam | Placebo | Midazolam | Total
Number analyzed (Participants) | 303 | 59 | 69 | 431
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (12.09) | 60.8 (12.08) | 61.5 (14.03) | 62.3 (12.41)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 154 | 32 | 36 | 222
  ≥65 years | 149 | 27 | 33 | 209
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 35 | 34 | 233
  Male | 139 | 24 | 35 | 198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 0 | 0 | 8
  Not Hispanic or Latino | 295 | 59 | 69 | 423
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 3 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 33 | 10 | 19 | 62
  White | 263 | 46 | 49 | 358
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 303 | 59 | 69 | 431
Height [Mean (Standard Deviation); unit: cm] | 168.6 (9.5) | 167.1 (10.0) | 170.0 (9.87) | 168.6 (9.64)
Weight [Mean (Standard Deviation); unit: kg] | 80.9 (20.21) | 77.7 (21.17) | 83.0 (22.10) | 80.8 (20.66)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (6.39) | 27.9 (7.09) | 28.0 (5.79) | 28.3 (6.39)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Successful Procedure
Description: Success of Procedure measured by completion of bronchoscopy, no requirement for an alternative rescue sedative medication and no requirement for more than 5 doses of study medication within any 15 minute period in the blinded arms (remimazolam/placebo) or no requirement for more than 3 doses within any 12 minute window in the open-label midazolam arm.
Time Frame: From first dose of study drug to removal of bronchoscope (average time not known)
Population: All patients who were randomized and were analyzed as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Remimazolam | Placebo | Midazolam
Number analyzed (Participants) | 310 | 63 | 73
Participants | 250 | 3 | 24
Statistical Analysis 1: Comparison: Remimazolam vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Rates = 0.7588, 95% CI 2-sided [0.6903 to 0.8274]

2. Secondary Outcome: Time to Start of Procedure
Description: The time from the first dose of study drug until bronchoscope insertion on Day 1
Time Frame: From first dose of study drug until insertion of the bronchoscope
Population: All patients who were randomized and were analyzed as randomized.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Remimazolam | Placebo | Midazolam
Number analyzed (Participants) | 310 | 63 | 73
minutes | 4.1 [4.0 to 4.8] | 17.0 [16.0 to 17.5] | 15.5 [13.8 to 16.7]

3. Secondary Outcome: Time to Fully Alert
Description: The time to fully alert defined as time to first of 3 consecutive Modified Observer's Assessment of Alertness and Sedation (MOAA/S) scores after the end of the bronchoscopy procedure (bronchoscope out).
  MOAA/S scores: 5 = Responds readily to name spoken in normal tone [alert], 4 =Lethargic response to name spoken in normal tone, 3 = Responds only after name is called loudly and/or repeatedly, 2 = Responds only after mild prodding or shaking, 1 = Responds only after painful trapezius squeeze, 0 = Does not respond to painful trapezius squeeze.
  MOAA/S scores were assessed by the investigators.
Time Frame: From the last dose of study drug or rescue sedative AND from end of bronchoscopy until the patient has recovered to fully alert
Population: Patients who do not reach the endpoint are censored at last MOAAS
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Remimazolam | Placebo | Midazolam
Number analyzed (Participants) | 302 | 60 | 68
minutes
  After last dose of study drug or rescue sedative | 11.6 [10.0 to 12.8] | 20.0 [15.3 to 31.0] | 18.0 [15.0 to 20.1]
  After bronchoscope out | 6.0 [5.2 to 7.1] | 13.6 [8.1 to 24.0] | 12.0 [5.0 to 15.0]

4. Secondary Outcome: Time to Ready for Discharge
Description: Time from the last dose of study drug or rescue sedative and from the end of bronchoscopy until discharge (defined as the ability to walk unassisted)
Time Frame: After the last dose of study drug AND after the end of the bronchoscopy, until discharge
Population: Patients who do not reach the endpoint are censored at last MOAAS
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Remimazolam | Placebo | Midazolam
Number analyzed (Participants) | 302 | 60 | 68
minutes
  after last dose of study drug or rescue sedative | 64.8 [62.0 to 68.5] | 93.0 [75.0 to 107.0] | 70.0 [67.0 to 87.0]
  After bronchoscope out | 60.0 [57.0 to 63.0] | 81.0 [70.0 to 100.0] | 66.0 [62.0 to 72.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events were collected from Day 1 until end of Follow-Up (Day 4 [+3/-1 days]). TEAEs were followed-up until events were resolved, became stable or could be explained by another known cause(s)
Description: Total number of participants affected with Other (Not Including Serious) Adverse Events represents any participant in the trial with a TEAE. The number of participants with Preferred Term (PT)TEAEs represents participants with non-serious TEAEs reported with a threshold of 5% in any of the arms
Arm/Group | Remimazolam | Placebo | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/303 | 0/59 | 0/69
Serious Adverse Events (participants affected / at risk) | 17/303 | 4/59 | 0/69
Other Adverse Events (participants affected / at risk) | 268/303 | 52/59 | 63/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remimazolam (N=303) | Placebo (N=59) | Midazolam (N=69)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atrial fibrillation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atrial tachycardia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bradycardia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remimazolam (N=303) | Placebo (N=59) | Midazolam (N=69)
Hypotension (Vascular disorders) | 99 | 28 | 23
Hypertension (Vascular disorders) | 85 | 9 | 19
Diastolic hypertension (Vascular disorders) | 77 | 15 | 16
Systolic hypertension (Vascular disorders) | 67 | 13 | 17
Diastolic hypotension (Vascular disorders) | 41 | 17 | 16
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 64 | 11 | 13
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 4
Respiratory rate increased (Investigations) | 43 | 6 | 10
Bradycardia (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 30 days prior to submission of communications, sponsor shall review and comment on the communications. Sponsor shall have the right to require institution and investigator to remove specifically identified confidential information and to delay the proposed publication an additional 45 days to enable sponsor to seek patent protection.

DOCUMENTS (2):
  • Study Protocol (2016-03-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT02296892/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT02296892/SAP_001.pdf